CLINICAL TRIAL: NCT04477031
Title: Verification of the Safety of Normal Food Before a Cerebral Arteriography
Acronym: VIANAC
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0396
Record Dates: First submitted 2020-07-10; First posted 2020-07-20 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Angiography
Keywords: Fasting; non fasting; cerebral angiography; nausea; vomiting
MeSH Terms: conditions — Fasting; Nausea; Vomiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Fasting is currently required before elective cerebral angiography, despite numerous arguments against fasting (kidney toxicity, vasovagal reaction, discomfort) and seams unusefull regarding it's main goal : reducing nausea and vomiting. The investigators propose to assess frequency of nausea and vomiting among patients having taken their breakfast at home before day care angiography.

The investigators hypothesise that less than 1% of non fasting patients will suffer of vomitint.

DETAILED DESCRIPTION:
Fasting is currently required before elective cerebral angiography, despite numerous arguments against fasting (kidney toxicity, vasovagal reaction, discomfort) and seams unusefull regarding it's main goal : reducing nausea and vomiting. The investigators propose to assess frequency of nausea and vomiting among patients having taken their breakfast at home before day care angiography.

The investigators hypothesise that less than 1% of non fasting patients will suffer of vomitint.

ELIGIBILITY:
Inclusion Criteria:

* Adult,
* non fasting,
* day care hosptilalisation

Exclusion Criteria:

* Childs,
* pregnancy,
* parenteral nutrition,
* nausea,
* vomiting before arteriography,
* arteriography under general anesthesia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients benefiting from a cerebral arteriography, within the UMCA of the North Laënnec Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 677 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
frequency of vomiting during arteriographic procedure | fifteen minutes
  The investigators check if there is vomiting or not during the examination noted by an electro radiology manipulator. Safety issue : Bronchus inhalation

SECONDARY OUTCOMES:
nausea | fifteen minutes
  The nausea will be evaluated using an analog visual scale (EVA) by an electro-radiology manipulator (MAR)at the exit of the intervention room

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Daumas-Duport, ph, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France